CLINICAL TRIAL: NCT02355457
Title: Biomarkers in Acute Cardiac Care
Acronym: BACC
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV4306
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Chest Pain
Keywords: troponin; myocardial infarction; acs; AMI; biomarker; BACC; high-sensitivity
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Biospecimen Retention: Samples With DNA — blood samples, white blood cells.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected acute myocardial infarction: Patients with recent onset symptoms suggesting acute myocardial infarction

SUMMARY:
The primary aim of the study is to investigate new cardiac biomarkers and algorithms to diagnose acute coronary syndrome in patients with suspected acute myocardial infarction.

DETAILED DESCRIPTION:
The primary aim of the study is to detect and evaluate new cardiac biomarkers, evaluate and improve acute coronary syndrome (ACS) risk scores, which takes into account clinical, gender specific, psycho-social and lifestyle-risk factors, protein patterns and genetic variability in addition to the classical risk factors with respect to the primary endpoint of acute myocardial infarction.

Secondary study aims are :

* To provide estimates for the incidence of ACS in patients presenting with recent onset chest pain;
* To provide accurate, quantifiable measures of precursors of ACS;
* DNA, RNA, cells, and serum/plasma for comprehensive genetic, gene expression and proteomic studies
* To explore the impact of ACS candidate genes on cardiovascular risk stratification by using genome-wide analyses and a biological systems approach;
* To explore proteins relevant for ACS;
* To allow the identification of new therapeutic targets;
* To evaluate the impact of socio-economic factors on ACS and CAD risk.

Patients will be followed up during the hospital stay. Afterwards a telephone follow-up will take place after 30 days, 6, 24 and 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms suggestive of acute myocardial infarction
* Ability to provide written informed consent in accordance with Good epidemiological Practice and local legislation
* Individuals at least 18 years old

Exclusion Criteria:

- Insufficient knowledge of the German language (able to understand and write the German language)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with suspected myocardial infarction in the emergency department or the chest pain unit of the University Hospital Hamburg-Eppendorf.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-07; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Acute myocardial infarction as index event | Months
  The primary endpoint of the study is acute myocardial infarction

SECONDARY OUTCOMES:
AMI, Mortality, heart failure and quality of life | Years
  The secondary endpoint of the study is mortality, heart failure, quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Neumann, MD, Principal Investigator — UHZ; Nils Sörensen, MD, Principal Investigator — UHZ
Locations (1):
- Department of Cardiology, University Heart Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Neumann JT, Sorensen NA, Schwemer T, Ojeda F, Bourry R, Sciacca V, Schaefer S, Waldeyer C, Sinning C, Renne T, Than M, Parsonage W, Wildi K, Makarova N, Schnabel RB, Landmesser U, Mueller C, Cullen L, Greenslade J, Zeller T, Blankenberg S, Karakas M, Westermann D. Diagnosis of Myocardial Infarction Using a High-Sensitivity Troponin I 1-Hour Algorithm. JAMA Cardiol. 2016 Jul 1;1(4):397-404. doi: 10.1001/jamacardio.2016.0695. PMID 27438315
- [Result] Neumann JT, Sorensen NA, Ojeda F, Schwemer T, Lehmacher J, Gonner S, Jarsetz N, Keller T, Schaefer S, Renne T, Landmesser U, Clemmensen P, Makarova N, Schnabel RB, Zeller T, Karakas M, Pickering JW, Than M, Parsonage W, Greenslade J, Cullen L, Westermann D, Blankenberg S. Immediate Rule-Out of Acute Myocardial Infarction Using Electrocardiogram and Baseline High-Sensitivity Troponin I. Clin Chem. 2017 Jan;63(1):394-402. doi: 10.1373/clinchem.2016.262659. Epub 2016 Nov 30. PMID 27903616
- [Derived] Haller PM, Schock A, Kellner C, Lehmacher J, Toprak B, Hartikainen TS, Kiss KM, Alhaou G, Peifer K, Twerenbold R, Zeller T, Westermann D, Neumann JT, Sorensen NA. Bedside echocardiography in patients with suspected acute myocardial infarction without ST elevation. Clin Res Cardiol. 2025 Aug 19. doi: 10.1007/s00392-025-02724-2. Online ahead of print. PMID 40828180
- [Derived] Thiebetaen N, Pickering JW, Kellner C, Haller PM, Lehmacher J, Toprak B, Twerenbold R, Sorensen NA, Pemberton C, Troughton R, Richards AM, Sharif S, Worster A, Than M, Kavsak PA, Neumann JT. A Common Algorithm for Cardiac Troponin to Rule Out and Rule in Acute Myocardial Infarction. Can J Cardiol. 2025 Jul;41(7):1351-1360. doi: 10.1016/j.cjca.2025.02.029. Epub 2025 Feb 26. PMID 40021054
- [Derived] Haller PM, Kellner C, Sorensen NA, Lehmacher J, Toprak B, Schock A, Hartikainen TS, Twerenbold R, Zeller T, Westermann D, Neumann JT. Long-term outcome of patients presenting with myocardial injury or myocardial infarction. Clin Res Cardiol. 2025 Jun;114(6):700-708. doi: 10.1007/s00392-023-02334-w. Epub 2023 Nov 20. PMID 37982865
- [Derived] Haller PM, Sorensen NA, Hartikainen TS, Gossling A, Lehmacher J, Toprak B, Twerenbold R, Richter J, Banko T, Korschid S, Schmidt J, Keller T, Zeller T, Blankenberg S, Westermann D, Neumann JT. Rising and Falling High-Sensitivity Cardiac Troponin in Diagnostic Algorithms for Patients With Suspected Myocardial Infarction. J Am Heart Assoc. 2023 May 16;12(10):e027166. doi: 10.1161/JAHA.122.027166. Epub 2023 May 9. PMID 37158171
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Aldous SJ, Allen BR, Apple FS, Babel H, Christenson RH, Cullen L, Di Carluccio E, Doudesis D, Ekelund U, Giannitsis E, Greenslade J, Inoue K, Jernberg T, Kavsak P, Keller T, Lee KK, Lindahl B, Lorenz T, Mahler SA, Mills NL, Mokhtari A, Parsonage W, Pickering JW, Pemberton CJ, Reich C, Richards AM, Sandoval Y, Than MP, Toprak B, Troughton RW, Worster A, Zeller T, Ziegler A, Blankenberg S; ARTEMIS study group. Personalized diagnosis in suspected myocardial infarction. Clin Res Cardiol. 2023 Sep;112(9):1288-1301. doi: 10.1007/s00392-023-02206-3. Epub 2023 May 2. PMID 37131096
- [Derived] von Haehling S, Muller-Hennessen M, Garfias-Veitl T, Gossling A, Neumann JT, Sorensen NA, Haller PM, Hartikainen T, Vollert JO, Mockel M, Blankenberg S, Westermann D, Giannitsis E. Role of Copeptin and hs-cTnT to Discriminate AHF from Uncomplicated NSTE-ACS with Baseline Elevated hs-cTnT-A Derivation and External Validation Study. Cells. 2023 Mar 31;12(7):1062. doi: 10.3390/cells12071062. PMID 37048135
- [Derived] Lehmacher J, Neumann JT, Sorensen NA, Gossling A, Schmidt SE, Zeller T, Blankenberg S, Westermann D, Clemmensen PM. Diagnostic performance of a device for acoustic heart sound analysis in patients with suspected myocardial infarction. Open Heart. 2023 Mar;10(1):e002090. doi: 10.1136/openhrt-2022-002090. PMID 36858602
- [Derived] Hartikainen TS, Gossling A, Sorensen NA, Lehmacher J, Neumann JT, Blankenberg S, Westermann D. Prognostic Implications of a Second Peak of High-Sensitivity Troponin T After Myocardial Infarction. Front Cardiovasc Med. 2022 Jan 31;8:780198. doi: 10.3389/fcvm.2021.780198. eCollection 2021. PMID 35174220
- [Derived] Neumann JT, Weimann J, Sorensen NA, Hartikainen TS, Haller PM, Lehmacher J, Brocks C, Tenhaeff S, Karakas M, Renne T, Blankenberg S, Zeller T, Westermann D. A Biomarker Model to Distinguish Types of Myocardial Infarction and Injury. J Am Coll Cardiol. 2021 Aug 24;78(8):781-790. doi: 10.1016/j.jacc.2021.06.027. PMID 34412811
- [Derived] Haller PM, Neumann JT, Sorensen NA, Hartikainen TS, Gossling A, Lehmacher J, Keller T, Zeller T, Blankenberg S, Westermann D. The association of anaemia and high-sensitivity cardiac troponin and its effect on diagnosing myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2021 Dec 18;10(10):1187-1196. doi: 10.1093/ehjacc/zuab066. PMID 34350455
- [Derived] Sorensen NA, Gossling A, Neumann JT, Hartikainen TS, Haller PM, Scharlemann L, Lehmacher J, Ziegler A, Blankenberg S, Zeller T, Nordholt G, Renne T, Westermann D. Diagnostic Validation of a High-Sensitivity Cardiac Troponin I Assay. Clin Chem. 2021 Sep 1;67(9):1230-1239. doi: 10.1093/clinchem/hvab070. PMID 34254126
- [Derived] Sorensen NA, Neumann JT, Ojeda F, Renne T, Karakas M, Blankenberg S, Westermann D, Zeller T. Differences in measurement of high-sensitivity troponin in an on-demand and batch-wise setting. Eur Heart J Acute Cardiovasc Care. 2021 May 11;10(3):302-309. doi: 10.1177/2048872620924198. Epub 2020 Jul 23. PMID 32700543
- [Derived] Neumann JT, Sorensen NA, Zeller T, Magaret CA, Barnes G, Rhyne RF, Peters C, Gossling A, Hartikainen TS, Haller PM, Lehmacher J, Schafer S, Januzzi JL, Westermann D. Application of a machine learning-driven, multibiomarker panel for prediction of incident cardiovascular events in patients with suspected myocardial infarction. Biomark Med. 2020 Jun;14(9):775-784. doi: 10.2217/bmm-2019-0584. Epub 2020 May 28. PMID 32462911
- [Derived] Haller PM, Boeddinghaus J, Neumann JT, Sorensen NA, Hartikainen TS, Gossling A, Nestelberger T, Twerenbold R, Lehmacher J, Keller T, Zeller T, Blankenberg S, Mueller C, Westermann D. Performance of the ESC 0/1-h and 0/3-h Algorithm for the Rapid Identification of Myocardial Infarction Without ST-Elevation in Patients With Diabetes. Diabetes Care. 2020 Feb;43(2):460-467. doi: 10.2337/dc19-1327. Epub 2019 Dec 16. PMID 31843947
- [Derived] Neumann JT, Twerenbold R, Ojeda F, Sorensen NA, Chapman AR, Shah ASV, Anand A, Boeddinghaus J, Nestelberger T, Badertscher P, Mokhtari A, Pickering JW, Troughton RW, Greenslade J, Parsonage W, Mueller-Hennessen M, Gori T, Jernberg T, Morris N, Liebetrau C, Hamm C, Katus HA, Munzel T, Landmesser U, Salomaa V, Iacoviello L, Ferrario MM, Giampaoli S, Kee F, Thorand B, Peters A, Borchini R, Jorgensen T, Soderberg S, Sans S, Tunstall-Pedoe H, Kuulasmaa K, Renne T, Lackner KJ, Worster A, Body R, Ekelund U, Kavsak PA, Keller T, Lindahl B, Wild P, Giannitsis E, Than M, Cullen LA, Mills NL, Mueller C, Zeller T, Westermann D, Blankenberg S; COMPASS-MI Study Group. Application of High-Sensitivity Troponin in Suspected Myocardial Infarction. N Engl J Med. 2019 Jun 27;380(26):2529-2540. doi: 10.1056/NEJMoa1803377. PMID 31242362
- [Derived] Sorensen NA, Nikorowitsch J, Neumann JT, Rubsamen N, Gossling A, Hartikainen TS, Blankenberg S, Westermann D, Zeller T, Karakas M. Predictive value of soluble urokinase-type plasminogen activator receptor for mortality in patients with suspected myocardial infarction. Clin Res Cardiol. 2019 Dec;108(12):1386-1393. doi: 10.1007/s00392-019-01475-1. Epub 2019 Apr 16. PMID 30989318
- [Derived] Neumann JT, Sorensen NA, Rubsamen N, Ojeda F, Schock A, Seddighizadeh P, Zeller T, Westermann D, Blankenberg S. Evaluation of a new ultra-sensitivity troponin I assay in patients with suspected myocardial infarction. Int J Cardiol. 2019 May 15;283:35-40. doi: 10.1016/j.ijcard.2018.12.001. Epub 2018 Dec 5. PMID 30528623
- [Derived] Boeddinghaus J, Nestelberger T, Twerenbold R, Neumann JT, Lindahl B, Giannitsis E, Sorensen NA, Badertscher P, Jann JE, Wussler D, Puelacher C, Rubini Gimenez M, Wildi K, Strebel I, Du Fay de Lavallaz J, Selman F, Sabti Z, Kozhuharov N, Potlukova E, Rentsch K, Miro O, Martin-Sanchez FJ, Morawiec B, Parenica J, Lohrmann J, Kloos W, Buser A, Geigy N, Keller DI, Osswald S, Reichlin T, Westermann D, Blankenberg S, Mueller C; APACE, BACC, and TRAPID-AMI Investigators. Impact of age on the performance of the ESC 0/1h-algorithms for early diagnosis of myocardial infarction. Eur Heart J. 2018 Nov 7;39(42):3780-3794. doi: 10.1093/eurheartj/ehy514. PMID 30169752
- [Derived] Kavsak PA, Neumann JT, Cullen L, Than M, Shortt C, Greenslade JH, Pickering JW, Ojeda F, Ma J, Clayton N, Sherbino J, Hill SA, McQueen M, Westermann D, Sorensen NA, Parsonage WA, Griffith L, Mehta SR, Devereaux PJ, Richards M, Troughton R, Pemberton C, Aldous S, Blankenberg S, Worster A. Clinical chemistry score versus high-sensitivity cardiac troponin I and T tests alone to identify patients at low or high risk for myocardial infarction or death at presentation to the emergency department. CMAJ. 2018 Aug 20;190(33):E974-E984. doi: 10.1503/cmaj.180144. PMID 30127037
- [Derived] Sorensen NA, Neumann JT, Ojeda F, Schafer S, Magnussen C, Keller T, Lackner KJ, Zeller T, Karakas M, Munzel T, Blankenberg S, Westermann D, Schnabel RB. Relations of Sex to Diagnosis and Outcomes in Acute Coronary Syndrome. J Am Heart Assoc. 2018 Mar 10;7(6):e007297. doi: 10.1161/JAHA.117.007297. PMID 29525782
- [Derived] Neumann JT, Sorensen NA, Rubsamen N, Ojeda F, Renne T, Qaderi V, Teltrop E, Kramer S, Quantius L, Zeller T, Karakas M, Blankenberg S, Westermann D. Discrimination of patients with type 2 myocardial infarction. Eur Heart J. 2017 Dec 14;38(47):3514-3520. doi: 10.1093/eurheartj/ehx457. PMID 29020401
- [Derived] Neumann JT, Sorensen NA, Ojeda F, Renne T, Schnabel RB, Zeller T, Karakas M, Blankenberg S, Westermann D. Early diagnosis of acute myocardial infarction using high-sensitivity troponin I. PLoS One. 2017 Mar 23;12(3):e0174288. doi: 10.1371/journal.pone.0174288. eCollection 2017. PMID 28333976
- [Derived] Sorensen NA, Neumann JT, Ojeda F, Schwemer T, Renne T, Schnabel RB, Zeller T, Karakas M, Blankenberg S, Westermann D. Challenging the 99th percentile: A lower troponin cutoff leads to low mortality of chest pain patients. Int J Cardiol. 2017 Apr 1;232:289-293. doi: 10.1016/j.ijcard.2016.12.167. Epub 2016 Dec 27. PMID 28087181